CLINICAL TRIAL: NCT03282292
Title: Central Venous Catheter Insertion Site and Catheter Colonization and Bloodstream Infection in Pediatric Cardiac Surgery
Brief Title: Central Venous Catheter Insertion Site and Colonization in Pediatric Cardiac Surgery
Acronym: PRECiSE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Co-PI responsible for study procedures moved to another hospital
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Marco Ranucci, Director Clinical Research, IRCCS Policlinico S. Donato
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PedCVC
Record Dates: First submitted 2017-09-12; First posted 2017-09-13 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Central Line-associated Bloodstream Infection (CLABSI); Central Venous Catheter Associated Bloodstream Infection; Heart; Surgery, Heart, Functional Disturbance as Result; Congenital Heart Disease; Newborn; Infection
MeSH Terms: conditions — Heart Defects, Congenital; Infections

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Jugular (Experimental): CVC insertion in the left or right internal jugular vein
  Interventions: Procedure: Internal jugular vein CVC insertion
- Femoral (Active Comparator): CVC insertion in the right or left femoral vein
  Interventions: Procedure: Internal jugular vein CVC insertion

INTERVENTIONS:
Procedure: Internal jugular vein CVC insertion — Double lumen CVC insertion in the internal jugular vein

SUMMARY:
Randomized controlled trial comparing femoral vs internal jugular insertion site of central venous catheters (CVC) in newborns and infants undergoing cardiac surgery. The experimental hypothesis is that the jugular insertion site is superior to the femoral in terms of catheter colonization.

DETAILED DESCRIPTION:
Background: in adult patients, the femoral site of insertion of CVC is notoriously at higher risk of colonization and central-line associated bloodstream infection (CLABSI) than other sites (jugular or subclavian). In pediatric patients, the femoral site is more commonly used than in adult patients, but there is no sound data on catheter colonization and CLABSI related to the insertion site. The experimental hypothesis of this randomized controlled trial (RCT) is that the jugular insertion site is less likely to induce catheter colonization and CLABSI than the femoral site.

Methods: 160 patients under 1 year and scheduled for cardiac surgery will be included in this RCT; patients will be randomly allocated to the jugular (J Group) or Femoral (F Group). CVC insertion will be performed by one out of three selected expert operators.

The primary endpoint is the catheter colonization based on identification of bacterial grow into the catheter at removal time; CLABSI and CRBSI rate based on the same bacterial identification into the catheter tip and in the blood culture performed in case of signs and symptoms of infection.

Secondary endpoints are mechanical complications defined as arterial puncture immediately identified during procedure, hemothorax and pneumothorax; and procedural difficulty during insertion defined as number of attempts, no guidewire progress, duration of the procedure (time from the completion of the sterile precaution barriers and the catheter fixation.

ELIGIBILITY:
Inclusion Criteria:

Planned cardiac surgery Age <1 year Eligibility for both insertion sites (jugular and femoral) for CVC Availability of at least one out of the three chosen expert operators

Exclusion Criteria:

Emergency surgery Known vascular anatomic anomalies Previous cardiac surgery in the last 6 months No expert operator availability Intensive Care unit before surgery Central venous catheter inside at the time of randomization

Withdraw criteria (only for the first endpoint):

Impossibility to placement catheter in the selected site.

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2019-09-12 (Actual); Study Completion 2019-10-12 (Actual)

PRIMARY OUTCOMES:
CVC colonization | 14 days
  CVC positive culture after removal
CRBSI | 14 days
  Positive CVC culture and blood stream infection for the same organism
CLABSI | More than 48 hours
  A laboratory-confirmed bloodstream infection where central line was in place for more than 48h.

SECONDARY OUTCOMES:
Mechanical complications | 1 day
  Defined as arterial puncture; hemothorax; pneumothorax
Procedural difficulty | 1 hour
  Defined by number of attempts; no guidewire progress

CONTACTS AND LOCATIONS:
Overall Officials: Marco Ranucci, MD, Study Director — IRCCS Policlinico S. Donato
Locations (1):
- IRCCS Policlinico S.Donato, San Donato Milanese, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes
The dataset will be made available at reasonable request
Supporting Information: Study Protocol, SAP
Time Frame: November 2017 - November 2020

REFERENCES:
- [Result] Collignon P, Soni N, Pearson I, Sorrell T, Woods P. Sepsis associated with central vein catheters in critically ill patients. Intensive Care Med. 1988;14(3):227-31. doi: 10.1007/BF00717995. PMID 3379183
- [Result] Pearson ML. Guideline for prevention of intravascular device-related infections. Part I. Intravascular device-related infections: an overview. The Hospital Infection Control Practices Advisory Committee. Am J Infect Control. 1996 Aug;24(4):262-77. doi: 10.1016/s0196-6553(96)90058-9. No abstract available. PMID 8870910
- [Result] de Jonge RC, Polderman KH, Gemke RJ. Central venous catheter use in the pediatric patient: mechanical and infectious complications. Pediatr Crit Care Med. 2005 May;6(3):329-39. doi: 10.1097/01.PCC.0000161074.94315.0A. PMID 15857534
- [Result] Karapinar B, Cura A. Complications of central venous catheterization in critically ill children. Pediatr Int. 2007 Oct;49(5):593-9. doi: 10.1111/j.1442-200X.2007.02407.x. PMID 17875082
- [Result] Casado-Flores J, Barja J, Martino R, Serrano A, Valdivielso A. Complications of central venous catheterization in critically ill children. Pediatr Crit Care Med. 2001 Jan;2(1):57-62. doi: 10.1097/00130478-200101000-00012. PMID 12797890
- [Result] Richards MJ, Edwards JR, Culver DH, Gaynes RP. Nosocomial infections in medical intensive care units in the United States. National Nosocomial Infections Surveillance System. Crit Care Med. 1999 May;27(5):887-92. doi: 10.1097/00003246-199905000-00020. PMID 10362409
- [Result] Stenzel JP, Green TP, Fuhrman BP, Carlson PE, Marchessault RP. Percutaneous femoral venous catheterizations: a prospective study of complications. J Pediatr. 1989 Mar;114(3):411-5. doi: 10.1016/s0022-3476(89)80559-1. PMID 2921683
- [Result] He C, Vieira R, Marin JR. Utility of Ultrasound Guidance for Central Venous Access in Children. Pediatr Emerg Care. 2017 May;33(5):359-362. doi: 10.1097/PEC.0000000000001124. PMID 28471906
- [Result] Sanchez Sanchez A, Giron Vallejo O, Ruiz-Pruneda R, Fernandez Ibieta M, Reyes Rios PY, Villamil V, Martinez-Castano I, Rojas Ticona J, Gimenez Aleixandre MC, Ruiz Jimenez JI. [Use of ultrasound for placement of central venous catheters in pediatrics: results of a national survey]. Cir Pediatr. 2017 Jan 25;30(1):9-16. Spanish. PMID 28585784
- [Derived] Silvetti S, Aloisio T, Cazzaniga A, Ranucci M. Jugular vs femoral vein for central venous catheterization in pediatric cardiac surgery (PRECiSE): study protocol for a randomized controlled trial. Trials. 2018 Jun 25;19(1):329. doi: 10.1186/s13063-018-2717-1. PMID 29941012